CLINICAL TRIAL: NCT05625347
Title: A Single-dose, Open-label, Multi-center, Randomized, 2-treatment Crossover Study to Compare the Pharmacokinetics, Pharmacodynamics, Safety and Tolerability of Acetylsalicylic Acid Powder for Oral Inhalation With Non-enteric-coated Chewable Aspirin in Adult Subjects With Obstructive or Restrictive Pulmonary Function
Brief Title: Study to Compare the Pharmacokinetics and Pharmacodynamics of ASA Powder for Oral Inhalation With Non-enteric-coated Chewable Aspirin in Adult Subjects With Obstructive or Restrictive Pulmonary Function
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: The pivotal study failed to meet the primary endpoint. Without a successful readout of the pivotal study, there was no longer a purpose for the supportive BORA-1A-C302 study.
Sponsor: Vectura, Inc. (Industry)
Collaborators: Syneos Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: BORA-1A-C302
Record Dates: First submitted 2022-11-01; First posted 2022-11-22 (Actual); Last update posted 2024-03-22 (Actual); Status verified 2024-03

CONDITIONS: Obstructive Pulmonary Function; Restrictive Pulmonary Function
Keywords: ASA; acetylsalicylic acid; cyclooxygenase-1 enzyme; COPD; oral inhalation; inhaled; myocardial Infarction
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Respiratory Aspiration; Myocardial Infarction

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm 1: I-ASA 100mg, then C-ASA 162mg tablet (Experimental): Treatment A: Single dose of 100 mg ASA powder for oral inhalation (I-ASA) via DPI.
  Treatment B: Single dose of 162 mg chewable non-enteric-coated Aspirin (C-ASA) tablets.
  Interventions: Drug: single dose (100 mg) of ASA; Drug: single dose (162 mg) of non-enteric-coated chewable aspirin tablets
- Arm 2: C-ASA 162mg tablet, then I-ASA 100mg (Experimental): Treatment A: Single dose of 162 mg chewable non-enteric-coated Aspirin (C-ASA)tablets.
  Treatment B: Single dose of 100 mg ASA powder for oral inhalation (I-ASA) via DPI.
  Interventions: Drug: single dose (100 mg) of ASA; Drug: single dose (162 mg) of non-enteric-coated chewable aspirin tablets

INTERVENTIONS:
Drug: single dose (100 mg) of ASA — powder for oral inhalation via a Dry Powder Inhaler (DPI)
Drug: single dose (162 mg) of non-enteric-coated chewable aspirin tablets — orally administered

SUMMARY:
The goal of this clinical trial is to compare the pharmacokinetics (PK) pharmacodynamics (PD), safety and tolerability of acetylsalicylic acid powder for oral inhalation (I-ASA) with non-enteric-coated chewable aspirin (C-ASA) in adult subjects with obstructive or restrictive pulmonary function.

In the first treatment period, subjects will be randomized to receive either a single dose (100 mg) of I-ASA powder via a Dry Powder Inhaler (DPI) OR a single dose (162 mg) of C-ASA tablets. After a washout period, subjects will be crossed over to receive the other treatment in the second treatment period. All subjects will receive both treatments during the study. Each single dose treatment will be followed by up to 24 hours of serial post-dose PK, PD, and safety/tolerability assessments.

DETAILED DESCRIPTION:
Up to 16 adult males and females subjects are planned for enrollment in this study, to achieve a minimum of 10 subjects with evaluable PD/PK, safety, and tolerability data:

* 5 subjects with obstructive lung function [i.e., diagnosed with chronic obstructive pulmonary disease (COPD)]; and
* 5 subjects with restrictive lung function

ELIGIBILITY:
Inclusion Criteria:

All Cohorts

* Subjects must meet all of the following criteria to be included in the study:
* Male or female, ≥ 40 years of age.
* BMI >18.0 and <35.0 kg/m2 and body weight ≥50.0 kg for males and ≥45.0 kg for females.
* Clinically stable as determined by medical history, physical examination, vital signs, and clinical laboratory evaluation.
* Female subjects of non-childbearing potential must be: post-menopausal; or surgically sterile at least 3 months prior to first dosing.
* Sexually active female subjects of childbearing potential must be willing to use an acceptable contraceptive method throughout the study as detailed in protocol.
* Smoker (no more than 25 cigarettes or equivalent daily) or non-smoker.

Obstructive Pulmonary Function Cohort

* Subject with a smoking history of at least 10 pack-years.
* Subject with an established diagnosis of COPD at least 12 months prior to the screening visit AND confirmed at screening by spirometry, with a post bronchodilator FEV1 greater than 40% and equal to or less than 70% of the subject's normal predicted value and a post-bronchodilator FEV1 greater than 40% and equal to or less than 70% of the subject's normal predicted value and a post-bronchodilator FEV1/ FVC ratio < 0.70.
* Subject on stable uninterrupted maintenance COPD therapy for at least 3 months prior to screening as per SoC and without any history of moderate or severe exacerbations within 6 months prior to screening.
* Non-symptomatic subject on stable uninterrupted maintenance COPD therapy, such that, in the judgement of the Investigator, on the day of dosing in each period, it would be safe to withhold the morning dose of the maintenance treatment until 2 hours post-dose and to withhold PRN short acting rescue bronchodilators from 1 hour pre-dose until 2 hours post-dose.

Restrictive Pulmonary Function Cohort

* Subject with a history and documented prior diagnosis of underlying chronic respiratory or cardiac disease with restrictive pulmonary function as confirmed at the screening visit by:
* FEV1/FVC ≥ 0. 7 and
* FVC < LLN (or < 80% predicted) and
* TLC < 5th percentile predicted (or < 80% predicted) and
* DLCO ≤ 75% to ≥ 35% predicted
* Continued uninterrupted SoC therapy for underlying disease for at least 12 consecutive weeks immediately prior to screening.
* Stable patient, such that, in the judgement of the Investigator, on the day of dosing in each period, it would be safe to withhold the morning dose of the maintenance treatment until 2 hours post-dose and to withhold short acting rescue bronchodilators, if any, from 1 hour pre-dose until 2 hours post-dose.

Exclusion Criteria:

All Cohorts:

* Presence of clinically significant uncontrolled or unstable cardiovascular, pulmonary, hepatic, renal, endocrinological, hematological, immunologic, metabolic, psychological, neurological, or gastrointestinal disease.
* Any new clinically significant abnormal finding at physical examination at screening.
* Positive serology test results for HBsAg, HCV antibody, or HIV antigen and antibody, or TB test at screening.
* Positive pregnancy test or lactating female subject.
* Positive urine drug screen or alcohol breath test.
* Positive test for active COVID-19.
* Known allergic reactions, hypersensitivity or contraindications to ASA, ibuprofen, other NSAID, or other related drugs, or to any excipient in the formulation.
* Known lack of response (lack of effect) to aspirin in the past.
* Clinically significant ECG abnormalities or vital signs abnormalities at screening.
* Clinically significant abnormal laboratory parameters at screening
* Presence of active or latent tuberculosis.
* History of asthma, including childhood asthma, syndrome of asthma, rhinitis (including allergic rhinitis), nasal polyps, angioedema, urticaria, angioedema, or bronchospasm that in investigator's opinion is not suitable to participate in the study.
* Subject with current asthma defined as post-bronchodilator FEV1 > 12% increase AND >200 ml absolute increase from pre-bronchodilator values.
* History of non-trauma related hemorrhage.

Restrictive Pulmonary Function Cohort

* Subject had lung surgery, with lung removal, as the reason for restrictive pulmonary function.
* Subject receiving systemic corticosteroid treatment of prednisone > 10 mg/day or equivalent within 3 months of screening.
* Subject suffers from restrictive pulmonary function, co-existent with obstructive pulmonary function disease.
* Subject has baseline resting oxygen saturation of < 89% on room air.
* Subject in need of continuous oxygen use and/or prescribed long-term continuous home oxygen therapy.

Other Protocol defined I/E criteria that apply

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2023-03-11 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2023-06-30 (Actual)

PRIMARY OUTCOMES:
Peak plasma concentration of ASA (Cmax) | pre-dose and 24 hours post-dose
Area under the ASA plasma concentration versus time curve (AUC0-inf) | pre-dose and 24 hours post-dose
Area under the ASA plasma concentration versus time curve (AUC0-t) | pre-dose and 24 hours post-dose

SECONDARY OUTCOMES:
Tmax of plasma concentrations of ASA. | assessed up to 24 hours post-dose
Tmax of plasma concentrations of SA. | assessed up to 24 hours post-dose
Peak Plasma Concentration (Cmax) of SA. | minutes post-dose: 2, 5, 10, 20, 30, 45, 60, 120, 180, 240, 360, 480, 720
Area under the plasma concentration versus time curve (AUC0-inf) of SA. | minutes post-dose: 2, 5, 10, 20, 30, 45, 60, 120, 180, 240, 360, 480, 720
Area under the plasma concentration versus time curve (AUC0-t) of SA. | minutes post-dose: 2, 5, 10, 20, 30, 45, 60, 120, 180, 240, 360, 480, 720
Serum thromboxane B2 (TxB2) serum concentration - Area under the effect curve (AUEC) of the % Change from baseline (CFB) in serum TxB2 concentration (TxB2 suppression). | 24 hours post-dose
TxB2 serum concentration - AUEC of the % CFB in serum TxB2 concentration (TxB2 suppression). | 20 minutes post-dose
TxB2 serum concentration - AUEC of the % CFB in serum TxB2 concentration (TxB2 suppression) | 30 minutes post-dose
Proportion of subjects achieving significant inhibition of platelet aggregation (<550 Aspirin Reaction Units [ARU]) | 2 minutes
Time to significant reduction in platelet aggregation (<550 ARU) | assessed up to 24 hours post-dose
Time to half-maximal % inhibition (suppression) of serum TxB2 (ID-50). | assessed up to 24 hours post-dose
Time to maximum % inhibition of serum TxB2. | assessed up to 24 hours post-dose
Time to maximum inhibition of platelet aggregation, assessed by VerifyNow Aspirin test. | assessed up to 24 hours post-dose
Maximum % CFB in ARU assessed by VerifyNow tests. | assessed up to 24 hours post-dose
Maximum % CFB in urinary 11-dehydro-TxB2. | assessed up to 24 hours post-dose
Maximum % CFB in serum 6-keto-PGF1α levels. | assessed up to 24 hours post-dose
Incidence and frequency of adverse events | Screening through the 7-day follow-up period

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - Omega Research Orlando, LLC, Orlando, Florida
  - Clinical Site Partners, LLC CSP Orlando, Winter Park, Florida
  - Sinai Hospital, Baltimore, Maryland
  - Hassman Research Institute, Berlin, New Jersey

IPD SHARING:
Plan to Share IPD: No